CLINICAL TRIAL: NCT00378404
Title: A Phase I Trial of Docetaxel and Low-Dose Fractionated Radiation in the Treatment of Metastatic or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase I Trial of Docetaxel and Low-Dose Fractionated Radiation in the Treatment of Metastatic or Recurrent NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Susanne Arnold (Other)
Collaborators: Kentucky Lung Cancer Research Program (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-LUN-69-UKY
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Non-Small Cell Lung Cancer; Non-Small Cell; Lung Cancer; Docetaxel; Radiation; Metastatic; Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Docetaxel; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Docetaxel; Radiation: Radiation

INTERVENTIONS:
Drug: Docetaxel — 30 mg/m2 IV on days 1, 8, 15 every 28 days for 6 cycles
Radiation: Radiation — 50 - 80 cGy on days 1, 8, 15 every 28 days for 6 cycles

SUMMARY:
The purpose of this study is to assess the maximum tolerated dose of low-dose radiation in combination with Docetaxel in recurrent or metastatic non-small cell lung cancer for second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or greater.
* Histologically or cytologically proven non-small cell lung cancer that is either metastatic or recurrent and failed at least one prior platinum-based chemotherapeutic regimen.
* Patients who have recurred after previous surgery and/or radiation may participate in this trial.
* Patients may have had prior neoadjuvant or adjuvant therapy.
* Patients with known brain metastases are eligible for this clinical trial if their disease has been treated and they are clinically stable and documented by a stable or improved pretreatment CT or MRI scan of the brain to evaluate for CNS disease within 28 days prior to registration.
* Measurable OR non-measurable disease documented by CT, MRI, X-ray or nuclear exam (FDG-PET). Measurable or non-measurable disease must be present outside the area of surgical resection. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease.
* Progression after at least one prior platinum-based chemotherapy.
* Greater than 3 weeks since surgery and must have recovered from all associated toxicities at time of registration.
* ANC ≥ 1,500/µl and platelet count ≥ 100,000/µl obtained within 28 days prior to registration.
* Adequate hepatic function documented by a serum bilirubin ≤ 1.5 times institutional upper limit of normal and liver enzymes (SGOT or SGPT) ≤ 2.5 x the institutional upper limit of normal obtained within 28 days prior to registration.
* Patients requiring lung radiation must have an FEV1 of > 1000 liters obtained within 28 days prior to registration and must have pulmonary function tests with DLCO.
* Zubrod Performance Status of 0,1 or 2.

Exclusion Criteria:

* No prior single-agent, weekly Docetaxel chemotherapy.
* Peripheral neuropathy ≥ Grade 1.
* Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 5 years.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess the MTD of low-dose fractionated radiation in combination with Docetaxel in recurrent or metastatic non-small cell lung cancer in the second-line setting. | continuously through treatment

SECONDARY OUTCOMES:
Toxicity | continuously throughout treatment
To investigate in an exploratory manner, the association of p53, p21^waf1/cip1, bcl-xL, bcl-2 and bax markers in pre- and post-treatment biopsies with patient response and toxicity. | week 1

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: University of Kentucky Markey Cancer Center Clinical Trials Listing — http://markey.uky.edu/studysearch